CLINICAL TRIAL: NCT06116604
Title: Early Bowel Resection for Terminal Ileal Crohn's Disease - Exploring Patients' and Clinicians' Perspectives and Barriers to Implementation
Brief Title: Early Bowel Resection for Terminal Ileal Crohn's Disease
Acronym: E-BRIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Centre for Health and Related Research (Unknown); University of Sheffield (Other); Crohn's & Colitis UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: STH21927
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; terminal ileitis; ileocaecal Crohn's; ileocaecal resection; bowel resection; shared decision-making; qualitative interviews; discrete choice experiment
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicentre mixed -methods study is to understand the patient and clinician perspective on the ideal timing of an operation for Crohn's disease of the terminal ileum (last part of the small bowel). The main questions it aims to answer are:

* What factors influence patients' and clinicians' preferences with regards to the timing of the first bowel resection for isolated Crohn's disease of the terminal ileum?
* What are patients' and clinicians' views on 'early' bowel resection (as an alternative to medical therapy) in this context?
* What are the facilitators and barriers to implementation of early surgery in practice?

Participants will be patients with Crohn's disease of the terminal ileum and healthcare professionals involved in treating inflammatory bowel disease.

Healthcare professionals have previously been asked to participate in an interview to understand their views on the role of surgery for Crohn's disease of the terminal ileum. They will now be invited to participate in a choice exercise to understand how much weight they attribute to various factors and outcomes when choosing between surgery and medication for Crohn's disease of the terminal ileum.

Patients will be asked to participate in:

1. an interview about their treatment choices
2. a choice exercise to understand how much weight they attribute to various factors and outcomes when choosing between surgery and medication for Crohn's disease of the terminal ileum
3. a survey, for patients with a previous ileocaecal resection, assessing their experience of the operation

DETAILED DESCRIPTION:
Crohn's disease is localised to the terminal ileum/ileocaecum in a third of patients. Typical medical therapy for ileocaecal Crohn's involves steroids to induce remission, followed by escalation to immunosuppression and/or of biological therapies for refractory disease to maintain remission. Surgery may be considered late in this treatment pathway, when medical therapies have been exhausted or when complications of the disease process arise.

There is a growing body of evidence supporting surgery as a valid option earlier in the treatment pathway. Studies have shown that surgery and medical treatment produce equivalent short term quality of life scores, and that earlier bowel resection is more cost effective. There is also a reduced need for medical therapy and subsequent surgery in patients having an earlier operation compared to those on conventional medical therapy.

Despite the evidence, the concept of "early" surgery has not universally translated into clinical practice. The purpose of this study is to understand why through a mixed-methods study with clinicians and patients. The patient components will be multi-centre (involving up to 10 NHS sites across England and Wales). The aims will be to establish:

1. the views of clinicians and patients on early primary bowel resection as an alternative to escalation of medical therapy in the context of terminal ileal Crohn's disease
2. at what point in the treatment pathway surgery is seen as an acceptable option
3. the facilitators and barriers to implementing early surgery
4. patient and clinician treatment preferences for terminal ileal Crohn's disease and factors influencing their decision-making

This study consists of the following work packages:

1. Interviews with healthcare professionals with an interest in inflammatory bowel disease to explore their views on the role of surgery for terminal ileal Crohn's disease - this has already been completed
2. Interviews with patients with terminal ileal Crohn's disease to explore their views on treatment options including surgery for terminal ileal Crohn's disease
3. Survey of patients with previous terminal ileal Crohn's disease to assess their decision-regret
4. Discrete choice experiment with clinicians and patients to understand the weight attributed to different factors and outcomes when choosing between medical treatment and surgery for terminal ileal Crohn's disease

ELIGIBILITY:
1. Qualitative interviews with patients with terminal ileal (TI) Crohn's disease (CD)

   Inclusion Criteria:
   * Any patient ≥18 years of age, with CD currently or previously affecting the terminal ileum or ileocaecum (with or without involvement of the ascending colon). Where the patient also has concomitant CD affecting other sites, this should be L1-dominant disease (i.e. where treatment is predominantly being required for, or symptoms are predominantly being caused by, disease of the terminal ileum).

   AND

   -The diagnosis of TI CD should have been made in the ten years preceding the start of the study.

   AND

   -The patient should either currently be on steroid-sparing treatment for TI CD, or should have previously been on such treatment (to include enteral nutrition, immunomodulator therapy or biologics), or should have had an ileocolic resection or right hemicolectomy for TI CD.

   Exclusion Criteria:
   * Patients who have never been on any treatment for their TI CD or who have only ever had steroids as treatment (i.e. no other medical or surgical treatment)
   * Unable to communicate in English
2. Discrete choice experiment Inclusion and exclusion criteria for patient participants are as above in 1.

Eligibility criteria for healthcare professionals are as follows:

1. Consultant colorectal surgeon with an interest or expertise in IBD, or
2. Consultant gastroenterologist with an interest or expertise in IBD, or
3. IBD clinical nurse specialist (IBD CNS), or
4. any doctor (medical or surgical) undertaking a fellowship in IBD following achievement of their Certificate of Completion of Training, working in an NHS trust in any part of the UK.

3. Survey of patients with previous ileocaecal resection for CD

Inclusion criteria:

* Any patient who had their first ileocaecal or ileocolic resection for Crohn's disease of the TI (confirmed using the pathology report for the resected specimen) within 7 years of the launch of the study. Patients who subsequently require a redo ileocolic resection (such as for recurrence in the neo-terminal ileum) during the 7 year study time frame chosen can still be included, as long as their first resection was within the study period.
* Age 18 years and above
* Resection with primary anastomosis or with a stoma
* Elective, emergency and semi-elective operations.

Exclusion criteria:

1. Ileocaecal or ileocolic resection performed as an emergency operation for the first presentation of Crohn's disease (i.e. in someone not previously diagnosed with Crohn's)
2. Incidental diagnosis of Crohn's disease as a result of resection performed for an alternative pathology
3. Resection in the three months preceding the launch of the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with terminal ileal Crohn's disease (current or previous) Healthcare professionals with an interest or expertise in inflammatory bowel disease
Sampling Method: Probability Sample
Enrollment: 496 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Themes | Within 10 years of diagnosis
  Themes generated from analysis of patient interviews
Trade off preferences for treatments | Within 10 years of diagnosis
  Relative importance of attributes from the analysis of the discrete choice experiment
Patient preference for timing of resection | Within 7 years of operation
  Primary outcome for survey of patients with a previous ileocaecal resection
Decision-regret | Within 7 years of operation
  Primary outcome for survey of patients with a previous ileocaecal resection

SECONDARY OUTCOMES:
Correlation of decision-regret score with pre-operative treatment experiences, Shared-decision making, body image score, selected post-operative outcomes | Within 7 years of operation
  Secondary outcome for survey of patients with a previous ileocaecal resection

CONTACTS AND LOCATIONS:
Overall Officials: Steven Brown, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No